CLINICAL TRIAL: NCT03871777
Title: Dietary Intake of Inorganic Nitrate in Vegetarians and Omnivores and Its Impact on Blood Pressure, Resting Metabolic Rate and the Oral Microbiome
Brief Title: Dietary Nitrate Intake in Vegetarians and Omnivores
Acronym: NO3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Plymouth (Other)
Collaborators: University of the West of Scotland (Other)
Responsible Party: Principal Investigator, Raul Bescos, Lecturer, University of Plymouth
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 15/16-469
Record Dates: First submitted 2019-03-09; First posted 2019-03-12 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Blood Pressure
Keywords: nitrate; vegetarian; nitrite; oral microbiome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegetarians (Active Comparator): Healthy vegetarians (vegans and lacto-ovo vegetarians) 18 and 50 years formed this arm.
  Interventions: Other: Placebo mouthwash; Other: Chlorhexidine mouthwash
- Omnivores (Sham Comparator): Healthy omnivores with similar characteristics of vegetarians (age, body mass index, gender and physical activity levels) formed this arm
  Interventions: Other: Placebo mouthwash; Other: Chlorhexidine mouthwash

INTERVENTIONS:
Other: Placebo mouthwash — Participants received placebo mouthwash (ultrapure unflavoured water) with which they rinsed their mouth for one minute, twice a day for 7 days. Resting metabolic rate and blood pressure were measured on day eight. Additionally, blood and saliva samples were taken from all the participants. Dietary records of seven days were also collected in order to confirm the foods and portion sizes consumed, preparation methods, recipes and any brand names.
Other: Chlorhexidine mouthwash — After using placebo and complete all the physiological measurements, participants were given a further one-week supply of antibacterial mouthwash containing 0.2% chlorhexidine (Corsodyl, GlaxoSmithKline, UK), encouraged to rinse their mouth for one minute, twice a day for 7 more days. They returned to the laboratory in 7 days to repeat all measurements in the same order.

SUMMARY:
Vegetarian diets are commonly associated with lower blood pressure levels. This has been related to greater consumption of inorganic nitrate, since vegetables are the main source of this anion. Dietary nitrate is reduced to nitrite by commensal bacteria in the mouth, which in turn leads to increased circulatory nitrite availability. Nitrite can form nitric oxide by several pathways promoting a reduction in the vascular tone and lower blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Healthy vegetarians (vegans and ovo-lacto vegetarians) following this dietary pattern for at least a year.
* Health omnivores

Exclusion Criteria:

* Smokers
* Individuals taking any medications or recreational drugs.
* Individuals with pre-existing medical conditions such as hypertension, diabetes, dyslipidaemia or dental conditions (gingivitis).
* Individuals using mouthwash or tongue scrapes were excluded from this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2018-11-12 (Actual)

PRIMARY OUTCOMES:
Dietary nitrate intake | 7 days
  Macro- and micronutrient intake of seven-day food diaries were analysed using a nutritional analysis software programme (Microdiet, Downlee Systems, Chapel-en-le-Frith, UK). Nitrate content of vegetables was mainly obtained from the European Food Safety Authority and additional data for spinach and lettuce from the Food Standards Agency. Nitrate and total polyphenol figures were uploaded to the Microdiet database prior to analysis.
Concentration of nitrate and nitrite in plasma and saliva | 7 days
  Whole blood was collected into lithium-heparin tubes (BD Vacutainer®, Becton Dickinson, Plymouth, UK) and rapidly centrifuged at 4,000 rpm and 4°C for 10 minutes. The plasma was then separated, frozen at -80°C until further analyses of nitrate and nitrite were performed. Non-stimulated saliva (3 milliliters) was also collected into a sterile falcon tube and rapidly frozen at -80°C. Then, nitrate and nitrite were measured in plasma and saliva using ozone-based chemiluminescence.
Change in blood pressure | 7 days
  Systolic, diastolic and mean arterial blood pressure was measured following British Hypertension Guidelines. Three successive supine readings were taken using an oscillometric device (Connex ProBP 3400 Digital Blood Pressure Device, Welch Allyn UK Ltd.) with a one minute rest between readings. The second and third readings were averaged to determine mean clinic blood pressure.
Change in oral nitrate-reducing capacity | 7 days
  Nitrate-reducing capacity of oral bacteria was analysed to compare vegetarians and omnivores and treatments (placebo mouthwash vs antibacterial mouthwash). Participants were instructed to hold 10 milliliters of water containing sodium nitrate (80 μicromols) in their mouth for 5 minutes. The mouth rinse was collected into a Falcon sterile tube and centrifuged (4,500 rpm, 4°C) for 10 minutes. The supernatant was collected and stored at -80°C before measuring absolute nitrite concentration.
Change in Resting Energy Expenditure | 7 days
  Resting Energy Expenditure was analysed using indirect calorimetry after using the placebo mouthwash and antibacterial mouthwash
Change oral microbiome | 7 days
  bundance of oral bacteria was analysed using 16S ribosomal ribonucleic acid (rRNA) after using the placebo mouthwash and antibacterial mouthwash.
  Salivary DNA was extracted using a DNA kit (QIAamp® DNeasy Blood & Tissue Kit). Polymerase chain reaction (PCR) amplification of the 16S rRNA V1-2 region was carried out using universal 16S primers 27 F (5'-AGA GTT TGA TCM TGG CTC AG-3') and 338 R (5'-GCW GCC WCC CGT AGG WGT-3'). Single band PCR products were purified and quantified with Qubit 2.0 Fluorometer (Invitrogen, CA, USA). Sequencing was performed on an Ion Torrent Personal Genome Machine.
Change in blood biomarkers | 7 days
  Blood markers were analyzed to assess differences between vegetarians and omnivores to control for diabetes and dyslipidaemia and to analyse the effect of antibacterial mouthwash.
  Whole blood glucose and lactate was measured using a biochemistry analyser (YSI 2300 Stat Plus, YSI Life Sciences, USA). Total cholesterol, triglycerides, high density lipoproteins (HDL) and low density lipoproteins (LDL) were analysed with enzymatic methods using the Roche 702 spectrophotometric module of a Cobas 8000 analyser (Roche Diagnostics Ltd, UK)

CONTACTS AND LOCATIONS:
Overall Officials: Raul Bescos, PhD, Study Director — University of Plymouth
Locations (1):
- Laboratory of Nutrition, Exercise & Health, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be shared as requested